CLINICAL TRIAL: NCT07076771
Title: Impact of Serum Testosterone Level on Angiographic Complexity of Coronary Lesions in Premature Ischemic Egyptian Males
Brief Title: Serum Testosterone Level on Angiographic Complexity of Coronary Lesions in Premature Ischemic Egyptian Males
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Remon Saleh Adly, Lecturer of Cardiovascular, Faculty of Medicine, Sohag University, Sohag, Egypt., Sohag University
Other Study IDs: Soh-Med-25-5-9PD
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Testosterone; Angiographic Complexity; Coronary Lesion; Premature Ischemia; Males

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Significant coronary artery disease (CAD) group: Patients with significant coronary artery disease
  Interventions: Other: Coronary Angiography; Other: Syntax Score
- Non-significant coronary artery disease (CAD) group: Patients with non-significant coronary artery disease
  Interventions: Other: Coronary Angiography; Other: Syntax Score

INTERVENTIONS:
Other: Coronary Angiography — All angiographic procedures will be performed. Coronary artery disease will be defined as >70% stenosis in at least one major epicardial artery or >50% the left main coronary artery.
Other: Syntax Score — The angiographic complexity of coronary artery disease (CAD) will be assessed using the SYNTAX score.

SUMMARY:
This study aims to investigate the association between serum testosterone levels and the angiographic complexity of coronary artery lesions in male patients under 45 years of age presenting with premature ischemic heart disease.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains a leading cause of morbidity and mortality worldwide. While traditionally associated with older populations, there is a growing incidence of premature CAD.

Testosterone, the primary male sex hormone, exerts various physiological effects beyond its role in reproductive function. It influences muscle mass, fat distribution, insulin sensitivity, and vascular tone. Low testosterone levels have been associated with adverse metabolic profiles, including increased adiposity, dyslipidemia, and insulin resistance, all of which are established risk factors for atherosclerosis. Furthermore, testosterone deficiency has been linked to endothelial dysfunction, a critical early event in the development of atherosclerotic plaques.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged <45 years.
* Diagnosed with premature ischemic heart disease.
* Undergoing elective coronary angiography for suspected coronary artery disease (CAD) .

Exclusion Criteria:

* History of acute coronary syndrome within the preceding 3 months.
* Prior diagnosis of hypogonadism or history of testosterone replacement therapy or anabolic steroid use.
* Active neoplasm or history of chemotherapy.
* Known hepatic cirrhosis, chronic kidney disease, or end-stage renal disease.
* Use of medications known to affect sex hormone levels (e.g., spironolactone, ketoconazole).
* Endocrine disorders such as sickle cell anemia or celiac disease.

Max Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male patients diagnosed with premature ischemic heart disease.
Study Population: This prospective study will be conducted at Sohag University Hospitals after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Serum testosterone level | Immediately after angiography (Up to 1 hour)
  Serum testosterone level will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.